CLINICAL TRIAL: NCT00593918
Title: Innate Immunity and RSV Infection in Children
Brief Title: Innate Immunity and Respiratory Syncytial Virus (RSV) Infection in Children
Acronym: IIRI
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 7K08HL071742-05 (NIH)
Record Dates: First submitted 2008-01-03; First posted 2008-01-15 (Estimated); Results first posted 2010-05-13 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-09

CONDITIONS: Respiratory Syncytial Virus Infection
Keywords: RSV, asthma, innate immunity, gene, cytokines
MeSH Terms: conditions — Respiratory Syncytial Virus Infections; Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Nasal samples Supernatant from Peripheral mononuclear cell stimulation cultures DNA
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Toll-like Receptor 4 -2026/GG Genotype: Toll-like Receptor 4 (TLR4) -2026/GG Genotype of interest hypothesized to be associated with less inflammation during Respiratory Syncytial virus (RSV) infection
- Toll-like Receptor 4 -2026/AG and AA Genotypes: Toll-like Receptor 4 (TLR4) -2026/AG and AA control genotypes hypothesized to be associated with more inflammation during respiratory syncytial virus (RSV) infection

SUMMARY:
In this project we will study the capacity for single nucleotide polymorphisms (SNP) in TLR4 gene to induce varying levels of inflammatory chemokine and cytokine production.

DETAILED DESCRIPTION:
Infection with RSV is the most common cause of respiratory tract illnesses (LRIs) in the first 3 years of life. There are significant social and health care costs associated with RSV-LRIs. More than 3% of US children are hospitalized each year due to RSV and 500 die annually. Several longitudinal studies have also suggested that children who have RSV-LRIs are at substantially increased risk of developing asthma in the first 3 years after infection and bronchial hyperresponsiveness (BHR) many years after the primary infection. Mechanisms involved in RSV disease are not well understood. Recent reports suggest that RSV may initiate the innate immune response through the pattern recognition receptor, Toll like receptor-4 (TLR4). In this project we will study the capacity for single nucleotide polymorphisms (SNP) in TLR4 gene to induce varying levels of inflammatory chemokine and cytokine production. It has been suggested that such a mechanism may result in altered immune responses to RSV infection and different clinical outcomes. This research has direct application to improving our understanding of bronchiolitis in early childhood, particularly those factors that influence severity of the disease, and may have implications for possible therapy of patients with bronchiolitis in the future.

ELIGIBILITY:
Inclusion Criteria:

1. Parental or sibling history of asthma.
2. Child must be less than 24 months of age.
3. Presence of viral upper or lower respiratory tract symptoms.

Exclusion Criteria:

1. History of recurrent wheezing requiring systemic corticosteroids.
2. Prior history of lung disease.
3. Birth < 36 weeks gestation.
4. Immunodeficiency
5. Treatment with ribavirin, systemic or inhaled corticosteroids during the RSV infection.
6. Congenital heart disease.
7. No history of parental or sibling asthma.
8. Less than 48 hour or more than 5 day duration of viral URI symptoms since the peak symptoms from RSV would be expected to occur from 2-5 days into course of infection.

Max Age: 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children who present with viral upper respiratory infections or bronchiolitis to their primary care physician. Upon consent, children willl have cheek samples for genotyping and nasal secretion samples to determine RSV infection.
Sampling Method: Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2003-11; Primary Completion 2008-05 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theresa W. Guilbert, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin-Madison, Madison, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study details planned during the first 4 months of the study. Recruitment period began during the RSV seasons from November to May each year from 2003-2008 in medical clinics.
Pre-assignment Details: Patients were enrolled if they met the enrollment criteria
Groups:
- Toll-like Receptor 4 GG Genotype: Toll-like Receptor 4 (TLR4) -2026/GG gentoype hypothesized to be associated with less inflammation during Respiratory syncytial virus (RSV) infection
- Toll-like Receptor 4 AG/AA Genotypes: Toll-like Receptor 4 (TLR4) -2026/AG and AA control genotypes hypothesized to be associated with more inflammation during Respiratory syncytial virus (RSV) infection
Period: Overall Study
Arm/Group | Toll-like Receptor 4 GG Genotype | Toll-like Receptor 4 AG/AA Genotypes
Started | 17 (Number of children with Toll-like Receptor 4 (TLR4) -2026/GG Genotype) | 74 (Number of children with Toll-like Receptor 4 (TLR4) -2026/AG and AA genotypes)
Completed | 12 (Some children did not come in for the blood draw at visit 2) | 50 (Some children did not come in for the blood draw at visit 2)
Not Completed | 5 | 24
Not completed — Withdrawal by Subject | 5 | 24

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Toll-like Receptor 4 GG Genotype | Toll-like Receptor 4 AG/AA Genotypes | Total
Number analyzed (Participants) | 17 | 74 | 91
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 17 | 74 | 91
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 0.78 (0.56) | 0.82 (0.54) | 0.82 (0.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 32 | 39
  Male | 10 | 42 | 52
Region of Enrollment [Number; unit: participants]
  United States | 17 | 74 | 91

OUTCOME MEASURES:

1. Primary Outcome: Nasal Interferon (IFN)-a2
Description: Interferon a2 was measured from nasal lavage samples by Luminex multiplex assay.
Time Frame: 1-5 days during acute illness (not after day 5 of illness)
Population: Analysis was per protocol based on the number of children enrolled by genotype and completed nasal washes at first visit.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Toll-like Receptor 4 GG Genotype | Toll-like Receptor 4 AG/AA Genotypes
Number analyzed (Participants) | 17 | 74
pg/ml | 10 (3) | 26 (31)
Statistical Analysis 1: Comparison: Toll-like Receptor 4 GG Genotype vs Toll-like Receptor 4 AG/AA Genotypes; Test type: Superiority or Other; p = 0.04, Mixed Models Analysis; A mixed random effects model was used both unadjusted and adjustment for relevant co-variates obtained from the literature

2. Primary Outcome: Percentage of Participants With Detected Nasal Interferon (IL)-2 Cytokine Expression
Description: IL-2 measured from nasal lavage samples by Luminex multiplex assay
Time Frame: 1-5 days during acute illness (not after day 5 of illness)
Measure: Number; unit: Percentage of Participants
Arm/Group | Toll-like Receptor 4 GG Genotype | Toll-like Receptor 4 AG/AA Genotypes
Number analyzed (Participants) | 12 | 50
Percentage of Participants | 0 | 44
Statistical Analysis 1: Comparison: Toll-like Receptor 4 GG Genotype vs Toll-like Receptor 4 AG/AA Genotypes; Test type: Superiority or Other; p = 0.14, Mixed Models Analysis — Analysis was per protocol based on the number of children enrolled by genotype and completed nasal washes at first visit; [statistical method as in outcome 1, analysis 1]

ADVERSE EVENTS:
Arm/Group | Toll-like Receptor 4 GG Genotype | Toll-like Receptor 4 AG/AA Genotypes
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/74
Other Adverse Events (participants affected / at risk) | 0/17 | 0/74

LIMITATIONS AND CAVEATS:
Subject withdraw before blood draw on second visit and small numbers recruited lead to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No